CLINICAL TRIAL: NCT07156292
Title: The Epidemiology Change From 2006 to 2022 of Infective Endocarditis in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, WANG-HUEI SHENG, National Taiwan University Hospital
Other Study IDs: 202309097RINB
Record Dates: First submitted 2025-04-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-04

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; epidemiology; 2006 to 2022
MeSH Terms: conditions — Endocarditis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study, not interventional — Observational study, not interventional

SUMMARY:
Infective endocarditis has long been one of the significant diseases causing death and disability worldwide. Its incidence has shown an increasing trend over the past few decades. Moreover, there seems to be significant variation in prevalence and epidemiology in different geographic regions and countries. This study aims to understand the trends and changes in the epidemiology of infective endocarditis in Taiwan from the 2006s to the present. Through a retrospective database analysis using the "Taiwan Healthcare System Integration Database," the goal is to improve the prognosis of infective endocarditis treatment in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were discharged from hospital or received an emergency diagnosis of infective endocarditis between January 1, 2006 and December 31, 2022

Exclusion Criteria:

* Patients without infective endocarditis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who were discharged from hospital or received an emergency diagnosis of infective endocarditis between January 1, 2006 and December 31, 2022
Sampling Method: Non-Probability Sample
Enrollment: 2247 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recent epidemiological trends and changes in infective endocarditis in Taiwan over the past decades | 2006 to 2022

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
local epidemiology in order
Supporting Information: Study Protocol